CLINICAL TRIAL: NCT05561179
Title: Hyaluronic Acid as a Novel Therapeutic Approach for Patients With GERD: a Single-center Study
Brief Title: Hyaluronic Acid in Patients With Gastroesophageal Reflux Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Principal Investigator, Carlos Robles-Medranda, Head of the Endoscopy Division, Instituto Ecuatoriano de Enfermedades Digestivas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IECED-09282022
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; hyaluronic acid; Esophageal Sphincter
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Hyaluronic Acid; Sodium Chloride; Control Groups

STUDY DESIGN:
Intervention Model Description: A non-blinded, single center, randomized prospective trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GERD + HA injections (Experimental): This group is comprised by patients with GERD, assessed previously through 24-Hour pH impedance test and esophageal manometry. The patients are submitted to HA injections at the lower esophageal level.
  Interventions: Procedure: Hyaluronic acid injection
- GERD without HA injections (Placebo Comparator): This group is comprised by patients with GERD assessed previously through 24-Hour pH impedance test and esophageal manometry. The patients are submitted to sodium chloride at the lower esophageal level.
  Interventions: Procedure: Sodium chloride injection (control group)

INTERVENTIONS:
Procedure: Hyaluronic acid injection — Patients with confirmed diagnosis of GERD will be treated with HA injections in the lower esophageal portion. HA + contrast will be injected in the 4 quadrants (4 cc/quadrant).
  The response to the treatment will be measured by improvement in health-related quality of life index, pH monitoring, and endoluminal functional lumen imaging probe (EndoFLIP). In addition, the patients will be clinically assessed for reflux symptoms.
  Arms: GERD + HA injections
Procedure: Sodium chloride injection (control group) — Patients with a confirmed diagnosis of GERD will be treated with sodium chloride injection in the lower esophageal portion. Sodium chloride + contrast will be injected in the 4 quadrants (4 cc/quadrant).
  The response to the treatment will be measured by improvement in health-related quality of life index, pH monitoring, and endoluminal functional lumen imaging probe (EndoFLIP). In addition, the patients will be clinically assessed for reflux symptoms.
  Arms: GERD without HA injections

SUMMARY:
Gastroesophageal reflux disease (GERD) remains one of the most common pathologies seen among gastroenterologists, surgeons, and primary care physicians. The high prevalence of this condition lead to further investigations in its prevention, diagnosis, and management. For the treatment of this chronic condition, improvement in quality of life and long-term durability should be considered.

Nowadays, proton pump inhibitors (PPIs) are considered the mainstay in the treatment of the patients with GERD; however, due to the increasing concern related to its safety in its long-term use and the over prescription of these drugs, new surgical and endoscopic interventions have emerged.

A local treatment based on injections of hyaluronic acid, a natural nonimmunogenic mucosal defense, in the lower esophageal mucosa is a tentative treatment option for these patients. Based on this, the investigators pursue to assess the effects of hyaluronic acid in gastroesophageal reflux control.

DETAILED DESCRIPTION:
GERD is one of the most common digestive pathologies, with a prevalence between 20% and 40% of adults. For the treatment of the disease, proton pump inhibitors (PPIs) have undoubtedly shown effective results; however, in around 30% of patients the complete resolution of symptoms fails.

For the latter, new therapeutic options should be considered. As a modern well-tolerated approach, and for local treatment, hyaluronic acid (HA) appeared to be an option for symptoms relief. HA is a glycosaminoglycan that acts as a natural defense for esophageal mucosa, able to organize the reticular structure as a filter to prevent the diffusion of high molecular substances. In addition, one of its remarkable features is the induction and control of epithelial cells turnover improving the re-epithelization process and the ulcer healing. In addition, hyaluronic acid compounds have shown no migration from the injection site in up to a three-year period.

Based on the above, the investigators aim to assess the effectiveness of hyaluronic acid in gastroesophageal reflux control, to considered it as an alternative effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old
* Patients with diagnosis of GERD (distal esophageal acid exposure time > 6% on 24hour ambulatory pH-impedance monitoring)
* Patients with abnormal distal esophageal acid exposure time (4%-6%) on 24-hour ambulatory pH-impedance monitoring
* Patients who authorized for endoscopic approach.

Exclusion Criteria:

* Pregnancy
* Any clinical condition which makes endoscopy inviable.
* Patients with severe anatomic conditions such as esophageal strictures, Barret´s esophagus, hiatal hernias.
* Previous esophageal surgery.
* Patients with a history of upper gastrointestinal neoplasia.
* Inability to provide informed consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Acid exposure to the distal esophagus after intervention | Up to 6 months
  The response to the therapy will be determined by the acid exposure to the distal esophagus, measured through pH monitoring and evaluated by 24-h acid exposure time (AET). AET is defined as the total time for which the pH in the distal esophagus is below 4 divided by the total duration of Multichannel Intraluminal Impedance (MII)-pH monitoring. It is expressed in percentages. AET of more than 4% is considered an abnormal distal esophageal acid exposure.
  The patients will be assessed at the beginning, one and six months after the procedure.
Assessment of esophageal transit and gastric emptying | Up to 1 month
  The assessment of gastrointestinal transit through barium x-ray (upper gastrointestinal series) to identify any post-procedural functional motility changes.
  The patients will be assessed one month after the procedure.
Change in health-related quality of life | up to 6 months
  Effect in the Gastroesophageal Reflux Disease Health-related quality of life through the Northwestern Esophageal Quality of Life (NEQOL) scale. NEQOL, a 14-item, single scale measure of Health-related quality of life (HRQOL), allows for rapid assessment in a clinical setting.
  The patients will be assessed at the beginning, and six months after the procedure.

SECONDARY OUTCOMES:
Evaluation of lower esophageal sphincter (LES) distensibility and pressure by EndoFLIP | Up to 1 month
  Based on pressure and distensibility evaluation of LES by EndoFLIP.
  The measure will be made at the beginning, and one month after the procedure.
Safety of HA injections in GERD | Up to 6 months
  Proportion of patients experiencing local adverse events related to the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MD FASGE, Principal Investigator — Instituto Ecuatoriano de Enfermedades Digestivas (IECED)
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas (IECED), Guayaquil, Guayas, Ecuador

REFERENCES:
- [Background] Katz PO, Dunbar KB, Schnoll-Sussman FH, Greer KB, Yadlapati R, Spechler SJ. ACG Clinical Guideline for the Diagnosis and Management of Gastroesophageal Reflux Disease. Am J Gastroenterol. 2022 Jan 1;117(1):27-56. doi: 10.14309/ajg.0000000000001538. PMID 34807007
- [Background] Martin K, Emil S, Bernard C, Gaied F, Blumenkrantz M, Laberge JM, Morinville V, Nguyen VH. Dextranomer hyaluronic acid copolymer effects on gastroesophageal junction. J Pediatr Gastroenterol Nutr. 2014 May;58(5):593-7. doi: 10.1097/MPG.0000000000000259. PMID 24345840
- [Background] Palmieri B, Merighi A, Corbascio D, Rottigni V, Fistetto G, Esposito A. Fixed combination of hyaluronic acid and chondroitin-sulphate oral formulation in a randomized double blind, placebo controlled study for the treatment of symptoms in patients with non-erosive gastroesophageal reflux. Eur Rev Med Pharmacol Sci. 2013 Dec;17(24):3272-8. PMID 24379055
- [Background] Pellegatta G, Mangiavillano B, Semeraro R, Auriemma F, Carlani E, Fugazza A, Vespa E, Repici A. The Effect of Hyaluronic Acid and Chondroitin Sulphate-Based Medical Device Combined with Acid Suppression in the Treatment of Atypical Symptoms in Gastroesophageal Reflux Disease. J Clin Med. 2022 Mar 29;11(7):1890. doi: 10.3390/jcm11071890. PMID 35407497
- [Background] Alshehri A, Emil S, Laberge JM, Elkady S, Blumenkrantz M, Mayrand S, Morinville V, Nguyen VH. Lower esophageal sphincter augmentation by endoscopic injection of dextranomer hyaluronic acid copolymer in a porcine gastroesophageal reflux disease model. J Pediatr Surg. 2014 Sep;49(9):1353-9. doi: 10.1016/j.jpedsurg.2014.02.088. PMID 25148736